CLINICAL TRIAL: NCT02263846
Title: Investigation of Sex Hormone Levels in Chinese Women With Invasive Breast Cancer
Status: Completed | Type: Observational
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Collaborators: Chinese Anti-Cancer Association (Other)
Responsible Party: Sponsor
Other Study IDs: CBCSG008
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Menopause; Estradiol; Follicle stimulating hormone
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Postmenopausal group: Patients at the age ≥ 60 years with more than one year of menopause, or patients having undergone bilateral oophorectomy.
- Premenopausal group: Patients with regular menses during recent 3 months and having never received luteinizing hormone-releasing hormone analogue therapy.

SUMMARY:
This study is to investigate sex hormones levels of Chinese patients with invasive breast cancer.The aim is to analyze biochemical monitoring results of premenopausal and postmenopausal patients to facilitate determination of menopausal status and propose clinical application.

DETAILED DESCRIPTION:
Follicle stimulating hormone (FSH), estradiol (E2) and luteinizing hormone (LH) can serve as indicators in the determination of menopausal status. NCCN clinical practice guidelines for breast cancer recommend detecting the levels of FSH and E2 for amenorrhea patients less than 60 years of age. But the detection method and the corresponding reference ranges indicating postmenopausal status are not mentioned. In addition, the reference limits vary a lot among different equipments and methods when it comes to diagnosis of menopause, thus it is difficult to set universal criteria. So in this study, four widely used methods and instruments in China are used to detect plasma levels of FSH, E2 and LN of premenopausal and postmenopausal patients. Instruments and methods must be one of the following four categories: microparticle chemiluminescent(Beckman),acridinium ester chemiluminescence (Siemens),acridinium ester chemiluminescence (Abbott) and electrochemiluminescence（Roche）.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer patients confirmed through pathology.
* For postmenopausal group: patients at the age ≥ 60 years with more than one year of menopause, or patients having undergone bilateral oophorectomy.
* For premenopausal group: patients with regular menses during recent 3 months and having never received luteinizing hormone-releasing hormone (LHRH) analogue therapy.
* Patients who meet the above criteria can be enrolled whether they have received anti-cancer treatment or not.

Exclusion Criteria:

* patients less than 60 years old who are amenorrhoeic but have not received bilateral oophorectomy or medical castration.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese women with invasive breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1183 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The capability of sex hormones to discriminate between pre- and postmenopausal women with invasive breast cancer measured by four widely used methods and instruments in China. | Two years
  Distribution characteristics of three hormones in pre- and postmenopausal patients are described with Kernel density estimation. Their discrimination capabilities are evaluated with operating characteristics (ROC) curve.

CONTACTS AND LOCATIONS:
Overall Officials: Santai Song, Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences

REFERENCES:
- [Background] Smith IE, Dowsett M, Yap YS, Walsh G, Lonning PE, Santen RJ, Hayes D. Adjuvant aromatase inhibitors for early breast cancer after chemotherapy-induced amenorrhoea: caution and suggested guidelines. J Clin Oncol. 2006 Jun 1;24(16):2444-7. doi: 10.1200/JCO.2005.05.3694. PMID 16735701